CLINICAL TRIAL: NCT04943705
Title: Evaluation of the Clinical Efficacy of Moxibustion With Regulating Yin and Yang in the Treatment of Menopausal Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hubei Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HubeiHTCM
Record Dates: First submitted 2021-06-13; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Obesity
Keywords: Menopausal Obesity; Yin and Yang Regulating Moxibustion; A Randomized Controlled Trial
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yin and Yang Regulating Moxibustion (Experimental): 1.The acupoints will be selected as Shenque and Mingmen.The location of the acupoints were based on the national GB/T 12346-2006 acupoints standard.Each treatment was 60min, once a week, Wenyang Yishen moxibustion and Peiyuan Guben moxibustion were performed alternately. Each patient received WenYang Yishen moxibustion and then Peiyuan Guben moxibustion for a total of 12 weeks of treatment and 12 weeks of follow-up at the end of the treatment. 2.The diet and exercise control implementation plan is as follows:Participants weighed ≤113.6 kg (250 lbs) and had a prescription diet of 1200-1499 kcal/day, including traditional foods, of which protein was about 15-20 kcal, fat was about 20-35%, and the rest came from carbohydrates. People weighing ≥113.6 kg are prescribed 1500-1800 kcal per day. They were also instructed to continue moderate-intensity physical activities (such as jogging, brisk walking) at least 5 days a week, at least 210 minutes a week, preferably ≥270 minutes a week。
  Interventions: Device: Yin and Yang Regulating Moxibustion
- Mild Moxibustion (Active Comparator): 1.The acupoints will be selected as Zhongwan, Guanyuan, Sanyinjiao (double).The location of the acupoints were based on the national GB/T 12346-2006 acupoints standard.Light one end of the moxa stick and hang it about 2-3cm above the skin, taking the patient's local skin redness and conscious warmth as the degree. Moxa-box moxibustion will be used for 20 minutes each treatment, once every other day, 3 times a week, for a total of 12 weeks of treatment, and 12 weeks of follow-up after the treatment. 2.Lifestyle modification:It will be performed as the same as the Yin and Yang Regulating Moxibustion group.
  Interventions: Device: Yin and Yang Regulating Moxibustion

INTERVENTIONS:
Device: Yin and Yang Regulating Moxibustion — Before making Wenyang Yishen moxibustion, the width and length of the patient's moxibustion site were evaluated by the same body measurement method. Take about 700g of fresh ground ginger with moderate dryness and wetness, and place it on the treatment towel to make a round cake with a diameter of about 20cm and a thickness of about 2.5cm. Spread 25g of moxa moxa with a diameter of about 18cm on top of ginger and light it. When the bottom temperature reaches about 37 degrees, the door can be placed on the patient's waist for treatment. According to the patient's tolerance, the temperature should be controlled at 43-45 degrees. It is better to replace the moxa biscuit every time when the moxa biscuit is burned for about 10 minutes. The patient's local skin has a slight redness and burning. The moxibustion time is 60 minutes. Peiyuan Guben moxibustion is centered on Shenque, and the operation is the same as that of WenYang and Yishen moxibustion.

SUMMARY:
This study is designed as a two-dummy randomized controlled trial to evaluate the safety and superiority of Yin and Yang regulating moxibustion in the treatment of menopausal obese patients.

DETAILED DESCRIPTION:
The study will be a multicenter, randomized, controlled trial, conducted from January 2021 to December 2022, including 216 menopausal obese patients who meet the inclusion criteria. The subjects will be randomly divided into 2 treatment groups: Yin and Yang regulating moxibustion group and mild moxibustion group. Each group of treatment will last for 12 weeks, with a follow-up period of 12 weeks. The main outcome indicator is waist circumference. The secondary outcome indicators include subjects related to obesity, TCM clinical syndrome score and modified Kupperman score, weight impact on quality of life scale (IWQOL-Lite), quality of life assessment health survey summary (SF-36). During the intervention period, adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnostic criteria for menopausal syndrome and obesity;
2. Patients with BMI≥25 and waist circumference≥80cm;
3. Female patients between 40-60 years old;
4. Have not taken any hormone drugs or weight loss related drugs in the past 3 months;
5. Sign the informed consent and voluntarily accept the intervention methods of this project.

Exclusion Criteria:

1. Unexplained vaginal bleeding, or unnatural menopause;
2. Have used hormone replacement therapy or other drugs related to this disease in the past 3 months;
3. Combined with serious organic diseases, endocrine diseases, heart, liver and kidney, and respiratory diseases;
4. Secondary obesity caused by hypothalamic lesions, hypothyroidism, glucocorticoid therapy, etc.;
5. Combined with organic uterine diseases, such as polycystic ovary syndrome, malignant tumors, severe cervical erosion, after total hysterectomy, etc.;
6. There are contraindications to moxibustion, such as moxibustion intolerance, skin allergies, scars, and other serious skin diseases;
7. Poor compliance and unable to adhere to treatment.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Obesity in female menopause
Enrollment: 216 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Waist circumference | Week 0, 4, 8, 12, 18and24.
  The change in waist circumference compared to the baseline.

SECONDARY OUTCOMES:
BMI(weight/height²) | Week 0, 4, 8, 12, 18and24.
  BMI (weight/height²) will be measured.
Weight(WG) | Week 0, 4, 8, 12, 18and24.
  Weight(WG) will be measured.
Hip circumference(HC) | Week 0, 4, 8, 12, 18and24.
  Hip circumference(HC) will be measured.
Waist-to-hip ratio(waist circumference/hip circumference) | Week 0, 4, 8, 12, 18and24.
  Waist-to-hip ratio(waist circumference/hip circumference) will be measured.
Body fat percentage(F percent) | Week 0, 4, 8, 12, 18and24.
  Body fat percentage(F percent) will be measured.
The syndrome score of Traditional Chinese Medicine | Week 0, 12and24.
  The syndrome score of Traditional Chinese Medicine will be adopted as the criterion of syndrome determination according to the diagnostic and therapeutic evaluation standard of simple obesity revised by the 5th National Obesity Research Conference in 1997. The minimum value is 0#the maximum value is 30. The lower the total score, the better of the outcome.
The impact of weight on quality of life (IWQOL)-Lite scale | Week 0, 12and24.
  The impact of weight on quality of life (IWQOL)- Lite scale will be measured. The minimum value is 31#the maximum value is 155. The lower the total score, the lighter the clinical symptoms of the patient.
Modified Kupperman score | Week 0, 12and24.
  The modified KMI score scale was used to evaluate the clinical symptoms of menopause before and after treatment.The minimum value is 0#the maximum value is 63. The lower the total score, the lighter the clinical symptoms of the patient.
The MOS Item Short from Health Survey（SF-36). | Week 0, 12and24.
  This scale is a universal health-related quality of life scale. The minimum value is 40#the maximum value is 147.The higher the comprehensive score, the better the quality of life.
Blood lipids: cholesterol (TC), triglycerides (TG), low-density lipoprotein (LDL-C), high-density lipoprotein (HDL-C). | Week 0 and 12.
  Compared with the baseline, the change value of this indicator.
Estrogen: estradiol (E2), serum follicle-forming hormone (FSH). | Week 0 and12.
  Compared with the baseline, the change value of this indicator.

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-Yu Zhou, professor, Principal Investigator — Hubei Hospital of Traditional Chinese Medicine
Locations (2):
- China (2):
  - Hubei Provincial Hospital of Traditional Chinese Medicine, Wuhan, Hubei
  - Zhong-Yu Zhou, Hubei

REFERENCES:
- [Derived] Yu B, Huang W, Zhang Y, Wang J, Xia C, Zhang Y, Xia H, Hu Y, Rao Y, Zhou Z. Efficacy and Safety of Moxibustion for Menopausal Obesity: A Multicentre, Randomized, Controlled Trial Protocol. Evid Based Complement Alternat Med. 2022 Aug 4;2022:9255017. doi: 10.1155/2022/9255017. eCollection 2022. PMID 35966744